CLINICAL TRIAL: NCT03789786
Title: Long-term Outcomes of Selective Dorsal Rhizotomy Among Individuals With Cerebral Palsy Compared to a Matched Control Group
Brief Title: Long-term Outcomes of Selective Dorsal Rhizotomy Among Individuals With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Michael H Schwartz, PhD, Director of Bioengineering Research, Gillette Children's Specialty Healthcare; Associate Professor of Orthopaedic Surgery, University of Minnesota - Twin Cities, Gillette Children's Specialty Healthcare
Other Study IDs: STUDY00002353
Record Dates: First submitted 2018-11-20; First posted 2018-12-31 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy
Keywords: Selective Dorsal Rhizotomy; Outcomes
MeSH Terms: conditions — Cerebral Palsy | interventions — Gait; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases (+SDR): Patients with cerebral palsy that underwent an SDR
  Interventions: Diagnostic Test: Gait and Motion Analysis; Diagnostic Test: Gross Motor Function Measure (GMFM); Behavioral: Surveys
- Controls (-SDR): Matched patients with cerebral palsy but did not undergo an SDR
  Interventions: Diagnostic Test: Gait and Motion Analysis; Diagnostic Test: Gross Motor Function Measure (GMFM); Behavioral: Surveys

INTERVENTIONS:
Diagnostic Test: Gait and Motion Analysis — Gait and motion analysis is comprised of 3-dimensional kinematics and kinetics, electromyography, energy expenditure, and physical exam (range of motion, strength, spasticity, etc.)
Diagnostic Test: Gross Motor Function Measure (GMFM) — Gross Motor Function Measure (GMFM) is an assessment used to evaluate gross motor function over time in individuals with cerebral palsy. The assessment is comprised of movement activities like standing, walking, running, and jumping
Behavioral: Surveys — Six surveys are used to assess function, activity, participation, pain, quality of life, and treatment history

SUMMARY:
Spasticity affects up to 80% of individuals diagnosed with cerebral palsy. Selective dorsal rhizotomy (SDR) is a surgical method used by some hospitals to permanently reduce spasticity in order to prevent further morbidities. Better understanding of the long-term outcomes of SDR is essential for clinicians and families. The results of this study will have direct clinical impact by equipping providers with the necessary information to counsel families during medical decision making.

DETAILED DESCRIPTION:
Spasticity affects up to 80% of individuals diagnosed with cerebral palsy. Excessive spasticity is thought to be uncomfortable, reduce function, cause gait deviations (e.g. equinus), and contribute toward musculoskeletal deformity and an elevated energy cost while walking. As such, SDR is a surgical method used by some hospitals to permanently reduce spasticity in order to prevent the aforementioned morbidities.

Treatment philosophies differ widely in regards to how aggressively to manage spasticity. Some centers (e.g. Gillette) aggressively treat spasticity early in life through a variety of measures such as SDR, intrathecal baclofen pumps, and botulinum toxin injections. Other centers (e.g. Shriners Hospitals for Children - Salt Lake City and Spokane) offer little in the way of spasticity reduction treatments.

There are several compelling reasons to conduct the proposed research study. First, emerging evidence suggests that the elimination of spasticity during childhood via SDR does not prevent contractures and only partially explains poor gross motor function, both previously thought to be clear outcomes of the surgery. Additionally, many of the longitudinal cohort studies that examined SDR outcomes have shown many outcome measures peak 1-3 years after surgery, and then decline toward baseline (i.e. pre-SDR) levels. Lastly, the quality of the SDR outcome literature is poor. Rarely are outcomes looked at in context of a proper control group. Either a control group is absent or comprised of typically developing children. This limits our ability to understand how patients with cerebral palsy may age without undergoing an SDR.

Better understanding of the long-term outcomes of SDR is essential for clinicians and families. The surgery, in general, is costly to families (time, expense, risk, etc.) and clinicians should have every confidence in the intended outcomes for any intervention.

ELIGIBILITY:
Inclusion Criteria for Controls (-SDR) and Cases (+SDR):

* Able to speak and read English
* Diagnosed with bilateral cerebral palsy (i.e. no hemiplegics)
* Minimum age of 21 years presently
* Had a baseline gait and motion analysis

Controls (-SDR):

* No SDR
* No history of intrathecal baclofen (ITB) pump implantation for > 1 year
* No ITB pump at time of long-term follow-up (explant > or = 6 months)
* No history of oral baclofen for > 1 year
* No oral baclofen use at time of long-term follow-up
* No more than 10 sessions on botulinum toxin, phenol, or alcohol injection

Cases (+SDR):

* History of SDR > 5 years ago
* Had a baseline gait analysis < or = 18 months before SDR

Exclusion Criteria:

* none

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Former/current patients at Gillette Children's Specialty Healthcare, Shriners Hospitals for Children - Salt Lake City, or Shriners Hospitals for Children - Spokane
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Three-dimensional gait and motion analysis | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Compare three-dimensional gait kinematics and kinetics across groups
Energy expenditure | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Compare energy expenditure across groups
Spasticity | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Compare spasticity, measured by Modified Ashworth Score (0 no increase in tone - 4 rigid in flexion or extension), across groups
Passive range of motion | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Compare passive range of motion, measured by lower extremity physical exam, across groups
Selective motor control | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Compare selective motor control (0 patterned movement - 2 complete isolated movement) across groups
Lower extremity strength | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Compare lower extremity strength, measured by the manual muscle test, across groups
Gross Motor Function Measure (GMFM-66) | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Assess function using portions of the GMFM-66 (0 low function - 100 high function) and compare across groups
Gillette Functional Assessment Questionnaire (Gillette FAQ) | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Assess function and activity using the Gillette FAQ (self-reported survey, 0 low function - 10 high function) and compare across groups
Functional Mobility Scale (FMS) | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Assess function and activity using the FMS (self-reported survey, 1 uses wheelchair - 6 independent) and compare across groups
Participation Enfranchisement survey | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Assess participation using the Participation Enfranchisement survey (self-reported survey, true/false) and compare across groups
Diener Satisfaction with Life Scale | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Assess satisfaction using the Diener Satisfaction with Life Scale (self-reported survey, 5 dissatisfied- 35 satisfied) and compare across groups
World Health Organization (WHO) Quality of Life Scale | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Assess satisfaction using the WHO Quality of Life Scale (self-reported survey, 0 low quality of life - 100 high quality of life) and compare across groups
Multiple Sclerosis Spasticity Scale (MSSS-88) | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Assess pain using portions of the MSSS-88 (self-reported survey, 21 not at all bothered - 84 extremely bothered) and compare across groups

SECONDARY OUTCOMES:
Change in gait and motion analysis | Baseline (qualifying exam for cases and controls) compared to long-term follow-up research visit (on average 10 years post-baseline)
  Compare change in gait kinematics and kinetics within groups and if the change is similar between groups
Incidence of prior surgery and anti-spastic treatments | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Incidence of prior surgery and anti-spastic treatments
Cost of prior surgery and anti-spastic treatments | Time of long-term follow-up research visit (on average 10 years post-baseline)
  Cost of prior surgery and anti-spastic treatments

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schwartz, PhD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (3):
- United States (3):
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Shriners Hospitals for Children - Salt Lake City, Salt Lake City, Utah
  - Shriners Hospitals for Childrens - Spokane, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munger ME, Chen BP, MacWilliams BA, McMulkin ML, Schwartz MH. Comparing the effects of two spasticity management strategies on the long-term outcomes of individuals with bilateral spastic cerebral palsy: a multicentre cohort study protocol. BMJ Open. 2019 Jun 20;9(6):e027486. doi: 10.1136/bmjopen-2018-027486. PMID 31227534